CLINICAL TRIAL: NCT03648164
Title: Development and Psychometric Test of CREATION Health Assessment Tool for College Students
Brief Title: CREATION Health Assessment Tool for College Students
Acronym: CHAT-CS
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1238224
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Health Behavior; Well Being
Keywords: well-being; health behavior; choice; rest; environment; activity; trust; interpersonal relationships; outlook; nutrition; survey; student; college; university
MeSH Terms: conditions — Health Behavior; Motor Activity; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CHAT-CS Survey — Students will complete a computer-based survey

SUMMARY:
CREATION Health encompasses eight whole-person care principles: Choice, Rest, Environment, Activity, Trust, Interpersonal-Relationships, Outlook, and Nutrition. An existing initial tool consisting of 74 items related to the eight CREATION Health principles and college students' wellbeing were generated by subject/methodology experts. To develop the CREATION Health Assessment Tool for College Students (CHAT-CS), this initial tool needs to be finalized through item reductions and validations in the population of college students.

DETAILED DESCRIPTION:
CREATION Health encompasses eight whole-person care principles: Choice, Rest, Environment, Activity, Trust, Interpersonal-Relationships, Outlook, and Nutrition.

Based on these principles, a health and wellness program, CREATION Health Wellness Program was developed. Since then various education/training plans using mind-body-spirit approaches have been implemented for different populations. Recently the Adventist Health System has plan to assess Adventist university students' health wellbeing and develop strategies to intervene and thus improve their overall wellbeing. However, literature review found that measures of these eight CREATION Health principles are often discrete and inconsistent. Therefore, there is an urgent need for a comprehensive, consistent assessment tool.

An existing initial tool consisting of 74 items related to the eight CREATION Health principles and college students' wellbeing were generated by subject/methodology experts. To develop the CREATION Health Assessment Tool for College Students (CHAT-CS), this initial tool needs to be finalized through item reductions and validations in the population of college students.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate college student
* Age 18 or more years
* Must be able to read and understand ENglish

Exclusion Criteria:

* Have previously taken the University Wellness Assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult undergraduate students in college/university
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Establish reliability using Cronbach's alpha | Through December, 2018
  Cronbach's (alpha) is a coefficient of reliability. The theoretical l value of the Cronbach's alpha varies from 0 to 1. A higher score indicates higher reliability.

SECONDARY OUTCOMES:
Item deduction | Through May, 2019
  * If an item is highly correlated with another item (item redundancy), consider removing one of the two items (correlation >.70)
  * If an item is not correlated (<.30) with other items, then consider eliminating this item
  * If an individual item has a weak loading on all factors (.39 or less), consider removing
  * If an item has a high loading (.40 or more) on multiple factors, consider modification or elimination

CONTACTS AND LOCATIONS:
Overall Officials: Hong Tao, PhD, Principal Investigator — AdventHealth
Locations (5):
- United States (5):
  - Oakwood University, Huntsville, Alabama
  - Andrews University, Berrien Springs, Michigan
  - Union College, Lincoln, Nebraska
  - Kettering College, Kettering, Ohio
  - Southern Adventist University, Collegedale, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johanson, G.A. and Brooks, G.P. (2010) Initial scare development sample size for pilot studies. Educational and Psychological Measurement, 70, 394-400.